CLINICAL TRIAL: NCT06512805
Title: Implementation Study of Intra-hospital Transfer of Pediatric Inpatients Based on the EPIS Model
Brief Title: Implementation Study of Intra-hospital Transfer of Pediatric Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CHFudanU1218
Record Dates: First submitted 2024-06-27; First posted 2024-07-22 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Implementation Science; Transportation of Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine transport group (Active Comparator): During the period from April 2024 to June 2024, pediatric patients transferred from the emergency department to the pediatric intensive care unit (PICU), and from the PICU to general wards will serve as the control group. They will undergo the hospital's current in-hospital transfer process.
  Interventions: Behavioral: Routine transport
- Post-guideline transfer group (Experimental): During the period from September 2024 to November 2024, pediatric patients transferred from the emergency department to the pediatric intensive care unit (PICU), and from the PICU to general wards will undergo the in-hospital transfer process based on the "Clinical Practice Guidelines for In-hospital Transfer of Pediatric Inpatients (2023 edition)."
  Interventions: Behavioral: Post-guideline transfer

INTERVENTIONS:
Behavioral: Routine transport — 1. Before the transfer of the patient:
     ① The doctor determines the destination of the patient based on the patient's condition and issues transfer orders.
     * The responsible nurse assesses the patient's consciousness, circulation, respiration, etc., and fills out the "Transfer Patient Handover Record" in the transferring department section.
       * The responsible nurse prepares the equipment, medications, and patient's belongings required for the transfer.
  2. During the transfer:
     Monitor the patient's vital signs.
  3. Upon arrival at the receiving department:
     * Place the patient with the receiving department nurse. ② Verbally hand over the patient's condition to the receiving department nurse and hand over the patient's belongings and medications.
       * The responsible nurse of the receiving department completes the remaining part of the "Transfer Patient Handover Record."
  Arms: Routine transport group
Behavioral: Post-guideline transfer — In the intervention group, nurses receive implementation strategies developed during the preparation phase. These strategies aim to modify the behavior of healthcare personnel through implementation, thereby conducting evidence-based (based on the guidelines) in-hospital transfer interventions for pediatric patients.The interventions received by pediatric patients are derived from the recommended practices evaluated for evidence availability in the guidelines. These include specific transfer procedures, the "Transfer Risk Level Classification Criteria," "Personnel Qualifications, Equipment, and Medications Allocation Based on Transfer Risk Level," "Transfer Preparation Checklist," and "Transfer Handover Checklist 2.0."
  Arms: Post-guideline transfer group

SUMMARY:
This study implemented the "Clinical Practice Guidelines for In-hospital Transfer of Pediatric Inpatients (2023 edition)" released by the research team in June 2023 in real clinical settings. It employed an effectiveness-implementation hybrid research design to evaluate the process and effects of the guidelines in clinical practice. The research objectives include the following aspects:

Identifying barriers to the implementation of the guidelines in clinical practice.

Constructing implementation strategies to facilitate the application of the guidelines based on identified barriers.

Evaluating the impact of implementation strategies on clinical healthcare personnel and the clinical environment.

Assessing the effect of in-hospital transfer of pediatric inpatients based on the guidelines on reducing adverse events related to in-hospital transfers and other clinical outcomes.

Participants will:

In the control group, healthcare personnel conduct transfers according to the routine management and working mode of the emergency department and pediatric intensive care unit (PICU).

In the intervention group, nurses receive implementation strategies developed during the preparation phase. These strategies are aimed at modifying the behavior of healthcare personnel through implementation, thereby conducting in-hospital transfers for pediatric patients based on the guidelines.

DETAILED DESCRIPTION:
The demand for in-hospital transfers is high, and their occurrence rate is frequent, making them an unavoidable routine in hospital settings due to emergency patients, postoperative patients, and those highly dependent on specialized medical equipment. Research statistics indicate that out of 371 patients admitted to the neonatal ward, there were 1402 transfers, while 506 emergency department patients accounted for 2715 in-hospital transfers. Additionally, 43.5% of patients in the intensive care unit required repeated transfers, with 45% of them needing two or more transfers. According to a systematic review by Haydar et al., adverse event rates during in-hospital pediatric transfers ranged from 0.11% to 75%, with the most common events being hypoxemia (13%-21%), hypotension (3.3%-37.5%), chest compressions (7.5%), dislodgement/accidental removal of catheters (3.8%), and interruption of vasopressor infusions (5%). Therefore, ensuring the safety of in-hospital transfers for pediatric patients is a crucial aspect of healthcare workers' responsibilities. Standardizing the in-hospital transfer process to minimize adverse events is vital for the well-being of pediatric patients.

Thus, this study focuses on in-hospital transfers of pediatric patients, aiming to identify current clinical issues and implement strategies based on the "Clinical Practice Guidelines for In-hospital Transfer of Pediatric Inpatients (2023 edition)." Conducted at the Children's Hospital affiliated with Fudan University, the research aims to develop implementation strategies and evaluate the impact of evidence and implementation strategies on pediatric inpatients, the evidence-based practice behavior of clinical healthcare personnel, and changes in the hospital organizational environment. The goal is to alter current clinical practices, standardize the in-hospital transfer process for pediatric patients, and further reduce adverse events associated with in-hospital transfers.

ELIGIBILITY:
Inclusion Criteria:

* Those who had worked in the study site for more than 1 year;

  * Those who can carry out intra-hospital transport independently;

    * Staff on duty during the study period

Exclusion Criteria:

* Those who have not obtained a practicing qualification certificate;

  * Refusal to participate in the study；

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The compliance of healthcare personnel with evidence-based practice. | Three months before and three months after the intervention
  The compliance of each review indicator = (Number of times the indicator was correctly executed / Total number of times the indicator was reviewed) * 100%.
Intra-hospital transfer time | Three months before and three months after the intervention
  The in-hospital transfer time = Time when the transfer team leaves the receiving department - Time when the transfer team leaves the transferring department.
Bedside handover time | Three months before and three months after the intervention
  Departure time of the transfer team from the receiving department - Start time of the handover.
Completeness of information handover | Three months before and three months after the intervention
  The ratio of completed items in the handover checklist to the total items in the handover checklist
Rate of adverse events during in-hospital transfers | Three months before and three months after the intervention
  Adverse event rate = Number of patients experiencing adverse events during transfer / Total number of patients transferred during the study period
Healthcare personnel's knowledge level of in-hospital transfers | One month before and one month after the intervention
  "In-hospital Transfer Knowledge Level Questionnaire for Healthcare Personnel"

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gu, Doctor, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No